CLINICAL TRIAL: NCT05302102
Title: Paretic-limb-only Plyometric Training Versus Volume-matched Double-limb Training for Ameliorating Balance Capability and Gait Symmetry in Adolescents With Unilateral Cerebral Palsy: A Comparative Study
Brief Title: Unilateral Versus Bilateral Lower-Limb Plyometric Training in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0019/0013
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: A prospective, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paretic-limb-only plyometric training group (Experimental): Participants in this group performed plyometric movements/exercises unilaterally using the paretic leg.
  Interventions: Other: Unilateral plyometric training
- Doule-limb plyometric training (Experimental): Participants in this group performed plyometric movements/exercises bilaterally through the paretic and non-paretic legs.
  Interventions: Other: Bilateral plyometric training
- Control group (Active Comparator): Participants in this group received the standard physical rehabilitation program.
  Interventions: Other: Standard physical therapy

INTERVENTIONS:
Other: Unilateral plyometric training — The paretic-limb-only plyometric training group received a plyometric exercise program performed unilaterally through the paretic leg only for 45 minutes, three times per week for 12 successive weeks. The training was conducted under close supervision of a licensed pediatric physical therapist according to safety performance guidelines defined by the American Academy of Pediatrics and the US National Strength and Conditioning Association.
  Arms: Paretic-limb-only plyometric training group
Other: Bilateral plyometric training — The double-limb plyometric training group received a plyometric exercise program performed bilaterally through the paretic and non-paretic legs for 45 minutes, three times per week for 12 successive weeks. The training was conducted under close supervision of a licensed pediatric physical therapist according to safety performance guidelines defined by the American Academy of Pediatrics and the US National Strength and Conditioning Association.
  Arms: Doule-limb plyometric training
Other: Standard physical therapy — The control group received the standard physical rehabilitation program conducted for 45 minutes, thrice a week for 12 consecutive weeks, and consisted of advanced balance training, gait training, postural and flexibility exercises, and strength training exercises.
  Arms: Control group

SUMMARY:
This study was set out to compare the effect of paretic-limb-only plyometric training versus double-limb training on balance capability and gait symmetry in adolescents with unilateral cerebral palsy (U-CP). Sixty-nine children with U-CP were randomly allocated to the paretic-limb-only plyometric training group (n = 23; performed plyometric movements/exercises unilaterally using the paretic leg only), the double-limb plyometric training group (n = 23; performed plyometric movements/exercises bilaterally through both lower legs), or the Control group (n =23, received standard rehabilitation plus SSC exercises). All groups were assessed for gait-symmetry and balance capability pre and post-treatment.

DETAILED DESCRIPTION:
Sixty-nine children with U-CP were recruited from the Physical Therapy Outpatient Clinic of College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, King Khalid Hospital, and a tertiary referral hospital, Al-Kharj, Saudi Arabia. Their age ranged between 12 and 18 years, were functioning at levels I or II according to the Gross Motor Function Classification System, and had spasticity level 1 or 1+ per the Modified Ashworth Scale. Children were excluded if they had fixed deformities, underwent neuromuscular or orthopedic surgery in the last 12 months, submitted to BOTOX injection in the past 6 months, had attentional neglect, and if they had cardiopulmonary problems preventing them from performing high-intense exercise training.

Outcome measures

* Gait-symmetry Indices: Gait symmetry indices (Spatial and temporal) were measured through the portable GAITRite system.
* Dynamic balance: The directional dynamic limit of stability (forward, backward, paretic, and non-paretic) and overall limit of stability were assessed using the Biodex balance system.

All groups were trained for 45 minutes, twice per week, for 12 successive weeks. The paretic-limb-only plyometric training group performed plyometric movements/exercises unilaterally using the paretic leg only. The double-limb plyometric training group performed plyometric movements/exercises bilaterally through both lower legs. The plyometric training program consisted of five unilateral and five bilateral lower limb plyometrics in the form of hopping/bounding/jumping activities. The plyometric training was preceded by a warm-up for 5 minutes and ended up with a 5-min cooldown. The control group received the standard rehabilitation program, which comprised advanced balance training, and gait training exercises, postural and flexibility exercises, strength training exercises.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral cerebral palsy
* Age 12-18 years
* Motor function level I or II according to the Gross Motor Function Classification System.
* Spasticity level 1 or 1+ according to the Modified Ashworth Scale

Exclusion Criteria:

* Structural deformities/contractures
* Musculoskeletal or neural surgery in the last year
* BOTOX injection in the last 6 months.
* Cardiopulmonary disorders that interfere with the ability to engage in exercise training.
* Perceptual and/or behavioral disorders.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Spatial gait symmetry | 2 months
  The spatial gait symmetry index was measured about the step length of the paretic and non-paretic leg through the portable GAITRite system. Lower scores indicate a more symmetrical pattern.
Temporal gait symmetry | 2 months
  The temporal gait symmetry index was measured about the single-limb support time of the paretic and non-paretic leg through the portable GAITRite system. Lower scores indicate a more symmetrical pattern
Limit of postural stability | 2 months
  The capacity to control and move the center-of-gravity in various directions across their base-of-support was assessed utilizing the Biodex balance system. Values are expressed as accuracy % and higher scores mean better balance capability.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No